CLINICAL TRIAL: NCT00665054
Title: Multi-centre, Randomized, Double-blind, Parallel, Placebo-controlled Clinical Study to Assess the Efficacy and Tolerability of Vardenafil and Its Influence on Self-esteem and Self Confidence in Subjects With Erectile Dysfunction.
Brief Title: BAY38-9456, 5/10/20mg, vs.Placebo in Erectile Dysfunction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11382
Record Dates: First submitted 2008-04-18; First posted 2008-04-23 (Estimated); Last update posted 2014-12-25 (Estimated); Status verified 2014-12

CONDITIONS: Erectile Dysfunction
Keywords: Vardenafil; Erectile dysfunction; SSES-E (sexual self-efficacy scale - erectile function)
MeSH Terms: conditions — Erectile Dysfunction | interventions — Vardenafil Dihydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Levitra (Vardenafil, BAY38-9456)
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levitra (Vardenafil, BAY38-9456) — 5, 10, or 20 mg Vardenafil tablets orally prior to sexual activity
  Arms: Arm 1
Drug: Placebo — Matching placebo tablets orally prior to sexual activity
  Arms: Arm 2

SUMMARY:
Purpose of the study is:- To assess the efficacy and tolerability of vardenafil in male subjects suffering from erectile dysfunction as compared to placebo- To assess the influence of vardenafil on the self-esteem and self-confidence of subjects suffering from erectile dysfunction following treatment with vardenafil as compared to placebo

ELIGIBILITY:
Inclusion Criteria:

* Men with heterosexual relationships aged 18 - 64 years suffering from ED for more than 6 months according to the NIH Consensus Statement (i.e. inability to attain and/or maintain penile erection sufficient for satisfactory sexual performance).
* At least 4 attempts at sexual intercourse (according to the question in the subject diary) on 4 separate days during the 4-week untreated baseline period. At least 50% of attempts during this period had to be unsuccessful according to the subject diary.

Exclusion Criteria:

* Presence of penile anatomical abnormalities (eg penile fibrosis or Peyronie's disease) that in the investigator's opinion would significantly impair sexual performance.
* Primary hypoactive sexual desire.-Spinal cord injury-History of surgical prostatectomy (transurethral interventions not excluded).
* Unstable angina pectoris.
* History of myocardial infarction, stroke or life-threatening arrhythmia within the prior 6 months.
* Uncontrolled atrial fibrillation/flutter at screening visit (ventricular response rate >100 BPM).

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2004-08; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
LOCF improved compared to baseline GAQ results at the end of the study | baseline versus visit 2 visit 5 or premature termination visit

SECONDARY OUTCOMES:
IIEF scores | visits 3, 4 and 5
OF, SD, IS scores in IIEF Questionnaire | visits 2, 3, 4, 5 or at premature termination visit
Scores of all individual questions on IIEF questionnaire | visits 2, 3, 4, 5 or at premature termination visit
Subject's diary response | baseline and after randomization per visit period
SSES-E scores | visits 2 and 5 or premature termination visit
Summary score from the responses to SSES-E | visits 2 and 5 or premature termination visit
Response scores and summary score from the responses to the SF-36 | visits 2 and 5 or premature termination visit

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (6):
- Turkey (Türkiye) (6):
  - Adana
  - Ankara
  - Antalya
  - Istanbul
  - Izmir
  - Samsun